CLINICAL TRIAL: NCT05409846
Title: Frequency of Fabry Disease in Portuguese Patients With Idiopathic Cardiomyopathies
Brief Title: Screening of Fabry Disease in Portuguese Patients With Idiopathic Cardiomyopathies
Acronym: F-CHECK
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Hospital Pedro Hispano (Other); Centro Hospitalar do Tâmega e Sousa, Hospital Padre Américo (Unknown); Hospital da Luz, Lisboa (Unknown); Centro Hospitalar De Trás-Os-Montes E Alto Douro, E.P.E. (Unknown); Centro Hospitalar Universitário Lisboa Norte, EPE., Hospital de Santa Maria (Unknown); Centro Hospitalar de Entre Douro e Vouga, E.P.E., Hospital São Sebastião (Unknown); Centro Hospitalar Universitário de Coimbra (Unknown); Centro Hospitalar de Vila Nova de Gaia e Espinho, E.P.E. (Unknown); Centro Hospitalar Universitário de Santo António (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: F-CHECK
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fabry Disease
Keywords: Idiopathic cardiomyopathies
MeSH Terms: conditions — Fabry Disease | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dry blood spot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: Idiopathic hypertrophic cardiomyopathy
  Interventions: Diagnostic Test: Alfa-galactosidase activity and genetic testing for Fabry diagnosis
- Group B: Idiopathic left ventricle hypertrophy
  Interventions: Diagnostic Test: Alfa-galactosidase activity and genetic testing for Fabry diagnosis
- Group C: Idiopathic burned-out hypertrophic cardiomyopathy
  Interventions: Diagnostic Test: Alfa-galactosidase activity and genetic testing for Fabry diagnosis
- Group D: Idiopathic dilated cardiomyopathy
  Interventions: Diagnostic Test: Alfa-galactosidase activity and genetic testing for Fabry diagnosis

INTERVENTIONS:
Diagnostic Test: Alfa-galactosidase activity and genetic testing for Fabry diagnosis — Dry blood spot analysis and blood sample (if necessary)

SUMMARY:
In Portugal, the prevalence of Fabry disease is largely unknown as recently has been stressed by the Portuguese hypertrophic cardiomyopathy registry investigators.

On the other hand, few data on Fabry screening protocols in patients with compromised ejection fraction including burned-out hypertrophic cardiomyopathy series have been published.

This project intends to perform screening of Fabry disease in patients with distinct cardiomyopathy phenotypes of unknown or dubious etiology and explore the less knew impact of the disease in other cardiac phenotypes.

ELIGIBILITY:
Inclusion Criteria:

Patients with heart disease diagnosed after the age of 30:

* unexplained hypertrophic cardiomyopathy (Group A)
* unexplained left ventricle hypertrophy confirmed in two different examinations using the same or different imaging methods (Group B)
* unexplained burned-out hypertrophic cardiomyopathy (Group C)
* unexplained dilated cardiomyopathy with evidence of late gadolinium enhancement involving the basal posterolateral wall segments (Group D)

Exclusion Criteria:

* previous exclusion of Fabry disease
* previous identified causal pathogenic/likely pathogenic genetic variant
* evidence of cardiomyopathy under the age of 30

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic cardiomyopathy patients
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Frequency of Fabry Disease in patients with idiopathic cardiomyopathies | 12 months
  Ratio of number of patients with Fabry Disease and total number of idiopathic cardiomyopathies patients

SECONDARY OUTCOMES:
Familiar screening of Fabry Disease | 12 months
  Number of relatives with Fabry Disease

CONTACTS AND LOCATIONS:
Overall Officials: Elisabete Martins, MD, PhD, Principal Investigator — Universidade do Porto
Locations (11):
- Portugal (11):
  - Centro Hospitalar Universitário de Coimbra, Coimbra
  - Hospital da Luz, Lisboa, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, EPE., Hospital de Santa Maria, Lisbon
  - Hospital Pedro Hispano (Unidade Local de Saúde Matosinhos), Matosinhos Municipality
  - Centro Hospitalar do Tâmega e Sousa, Hospital Padre Américo, Penafiel
  - Centro Hospitalar Universitário de Santo António, Porto
  - Centro Hospitalar Universitário São João, E.P.E., Porto
  - Faculty of Medicine (FMUP), Porto
  - Centro Hospitalar de Entre Douro e Vouga, E.P.E., Hospital São Sebastião, Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia e Espinho, E.P.E., Vila Nova de Gaia
  - Centro Hospitalar De Trás-Os-Montes E Alto Douro, E.P.E., Vila Real